CLINICAL TRIAL: NCT06655155
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase 2, Parallel-Group Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Efgartigimod PH20 SC in Adult Participants With Systemic Sclerosis
Brief Title: A Study to Assess the Efficacy and Safety of Efgartigimod PH20 SC in Adults With Systemic Sclerosis
Acronym: eSScape
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2317; 2024-514539-67-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod PH20 SC (Experimental): Participants receiving efgartigimod PH20 SC
  Interventions: Combination Product: Efgartigimod PH20 SC
- Placebo PH20 SC (Placebo Comparator): Participants receiving placebo PH20 SC
  Interventions: Other: Placebo PH20 SC

INTERVENTIONS:
Combination Product: Efgartigimod PH20 SC — Subcutaneous efgartigimod PH20 SC given by prefilled syringe
  Arms: Efgartigimod PH20 SC
Other: Placebo PH20 SC — Subcutaneous placebo PH20 SC given by prefilled syringe
  Arms: Placebo PH20 SC

SUMMARY:
The main purpose of this study is to evaluate the effect and safety of efgartigimod PH20 SC compared to placebo in adults with systemic sclerosis. The study consists of a screening period, a treatment period of up to 48 weeks and a safety follow-up period. After the screening period, eligible participants will be randomized in a 2:1 ratio to receive either efgartigimod PH20 SC or placebo. The total study duration can be up to approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Is aged ≥18 years and the local legal age of consent for clinical studies
* Has diffuse or limited SSc diagnosis and fulfills the 2013 ACR/EULAR classification criteria
* Has a positive antinuclear antibodies (ANA) test result at the central laboratory with titer of at least 1:160
* Has a Health Assessment Questionnaire-Disability Index (HAQ-DI) score of at least 0.5 OR a Patient Global Assessment (PGA) score of at least 3
* Has a modified Rodnan Skin Score (mRSS) score between 15 and 35
* The participant is anti-RNA polymerase III autoantibody negative at central laboratory and had the first non-Raynaud's phenomenon manifestation less than 5 years before screening or the participant is anti-RNA polymerase III autoantibody positive at central laboratory and had the first non-Raynaud's phenomenon manifestation less than 2 years before screening
* Has uninvolved or mildly thickened skin area in at least 1 injection site

Exclusion Criteria:

* Isolated anticentromere antibodies (ACA) seropositivity at the central laboratory
* Significant Pulmonary Arterial Hypertension
* Severe digital vasculopathy within the past 3 months
* Skin thickening due to scleroderma mimics or localized scleroderma
* Scleroderma renal crisis within the past 6 months of participating to the study
* Another rheumatic autoimmune disease, except for secondary Sjögren's syndrome or fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mRSS at week 24 | Up to 24 weeks
  The Modified Rodnan Skin Score is a scoring tool to assess skin thickness in 17 cutaneous sites across the body. Each site is rated on a semiquantitative score ranging from 0 (normal) to 3 (severe). The total score is the sum of the individual skin scores and can range from 0 to 51.

SECONDARY OUTCOMES:
Change from baseline in mRSS at week 48 | Up to 48 weeks
  The Modified Rodnan Skin Score is a scoring tool to assess skin thickness in 17 cutaneous sites across the body. Each site is rated on a semiquantitative score ranging from 0 (normal) to 3 (severe). The total score is the sum of the individual skin scores and can range from 0 to 51.
Incidence of treatment-emergent (serious) adverse events | Up to 55 weeks
Proportion of participants who improve in at least 2 or at least 3 of the 5 core items of CRISS-25 at weeks 24 and 48 and do not have worsening in >1 component and have no significant SSc-related event(s) | Up to 48 weeks
  Revised Composite Response Index in Systemic Sclerosis (CRISS-25) is a global composite outcome assessment that provides a holistic perspective of the disease. It includes 5 core items: the Modified Rodnan Skin Score, the Clinician's global assessment, the Forced Vital Capacity, the Patient global assessment, and the Health Assessment Questionnaire-Disability Index.
Change from baseline in HAQ-DI at weeks 24 and 48 | Up to 48 weeks
  Health Assessment Questionnaire-Disability Index is a tool to assess physical function and disability. It consists of 8 categories with each question scored from 0 (without any difficulty) to 3 (unable to do).
Change from baseline in PGA at weeks 24 and 48 | Up to 48 weeks
  Patient's Global Assessment is a tool that measures a participant's global evaluation of their overall health during the previous week using a 10-point numerical scale. The score varies between 0 (excellent overall health) and 10 (extremely poor overall health).
Change from baseline in CGA at weeks 24 and 48 | Up to 48 weeks
  Clinician's Global Assessment is a tool that measures a clinician's assessment of the overall health of a participant during the previous week using a 10-point numerical scale. The score varies between 0 (excellent overall health) and 10 (extremely poor overall health).
Annualized rate of decline in FVC (in mL) in participants with interstitial lung disease | Up to 48 weeks
  Forced Vital Capacity is a tool to assess lung function
Efgartigimod serum concentrations over time | Up to 48 weeks
Percent change from baseline in total IgG levels in serum over time | Up to 55 weeks
Incidence of anti-drug antibodies against efgartigimod in serum over time | Up to 55 weeks
Incidence of antibodies against rHuPH20 in plasma over time | Up to 55 weeks

CONTACTS AND LOCATIONS:
Locations (69):
- United States (9):
  - Arizona Arthritis and Rheumatology Associates, Phoenix, Arizona
  - UCLA Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - IRIS Research and Development LLC, Plantation, Florida
  - University of Illinois Health Outpatient Care Center, Chicago, Illinois
  - DelRicht Research, LLC, New Orleans, Louisiana
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Thomas Jefferson University, Columbia, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
- Argentina (7):
  - Aprillus Asistencia e Investigacion, Buenos Aires
  - Instituto de Investigación Clínica TyT, Buenos Aires
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Buenos Aires
  - Sanatorio Allende S.A., Córdoba
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán
  - Centro de Investigaciones Médicas Tucumán, San Miguel de Tucumán
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Brussel, Jette
- Bulgaria (2):
  - Medical Center Artmed OOD, Plovdiv
  - Diagnostic Consultative Center Convex EOOD, Sofia
- Chile (3):
  - BIOCINETIC Ltda, Santiago
  - Centro de Investigaciones Clinicas UC (CICUC), Santiago
  - Centro de especialidades médicas Vanguardia, Temuco
- Croatia (3):
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital of Split, Split
  - General Hospital Zadar, Zadar
- Revmatologicky Ustav, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU de Lille - Hopital Claude Huriez, Lille
  - CHU de Strasbourg - Hôpital de Hautepierre, Marseille
  - CHU de Montpellier- Hôpital Saint Eloi, Montpellier
  - AP-HP - Hôpital Cochin - Port-Royal, site Cochin, Paris
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Mühlenkreiskliniken - Johannes Wesling Klinikum Minden, Minden
  - Universitätsklinikum Tübingen, Tübingen
- Greece (3):
  - Olympion General Clinic, Pátrai
  - University General Hospital of Patras, Pátrai
  - Euromedica Kianous Stavros, Thessaloniki
- Pecsi Tudomanyegyetem, Klinika Kozpont, Bor, Nemikortani es Onkodermatologiai Klinika, Pécs, Hungary
- Italy (6):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipeda Hospital, Affiliate of Klaipeda University Hospital, Klaipėda
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (5):
  - Malopolskie Badania Kliniczne, Krakow
  - Zespol Poradni Specjalistycznych REUMED, Lublin
  - Twoja Przychodnia NCM, Nowa Sól
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Biogenes, Wroclaw
- Portugal (3):
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - ULS de Santa Maria,EPE - Hospital de Santa Maria, Lisbon
  - ULS de Gaia/Espinho, EPE - Unidade I, Vila Nova de Gaia
- The Alliance Medical Sciences Campus, San Juan, Puerto Rico
- Romania (2):
  - Sf.Maria Clinical Hospital, Bucharest
  - Dr I Cantacuzino Clinical Hospital, Bucharest
- Military Medical Academy, Belgrade, Serbia
- Spain (3):
  - Hospital Del Mar, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Corporacio Sanitaria Parc Tauli, Sabadell
- Switzerland (2):
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital, London
  - Luton and Dunstable University Hospital, Luton

IPD SHARING:
Plan to Share IPD: No